CLINICAL TRIAL: NCT07272447
Title: The Effect of Arm Message on the Success of Peripheral Intravenous Catheter Insertion in Breast Cancer Patients Undergoing Chemotherapy
Brief Title: Effect of Hand Message on Catheter Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Handan Eren, Associate Professor, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 224/187
Record Dates: First submitted 2025-07-07; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: vein visibility; breast cancer; peripheral catheter insertion
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): hand massage
  Interventions: Other: Hand massage
- control group (No Intervention): no intervention has applied

INTERVENTIONS:
Other: Hand massage — Classical hand massage that inclued effleurage, and petrisage.
  Arms: experimental group

SUMMARY:
This is a randomized controlled study to investigate the effect of arm message on the success of peripheral intravenous catheter insertion in breast cancer patients undergoing chemotherapy. There are two groups in our study (control group=30, experimental group=30). The investigator applied hand massage to patients in experimental group before peripheral intravenous catheter insertion. The investigators evaluated the succesfull peripheral catheter insertion time, anxiety level, and satisfaction level of the patients.

DETAILED DESCRIPTION:
Introduction: Peripheral intravenous catheter (PIVK) placement becomes difficult in patients diagnosed with breast cancer who receive chemotherapy because vein visibility decreases.

Objective: The aim of this study is to determine the effect of arm massage applied to patients diagnosed with breast cancer receiving chemotherapy on the success of peripheral intravenous catheter placement.

Method: The study will conducted in a randomized controlled experimental type in an outpatient chemotherapy unit of a hospital.The sample of the study will consist of 60 patients who met the inclusion criteria (experimental group = 30, control group = 30). Patients in the experimental group will receive arm massage before peripheral intravenous catheter placement, while patients in the control group will receive no intervention. The time to successful catheter placement, patient anxiety, and satisfaction levels regarding the procedure will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as breast cancer,
* having had the first course of chemotherapy,
* patients who has 1,2 and 3 vein degree

Exclusion Criteria:

* More than 2 unsuccessful attempts at PICK placement,
* The individual wants to leave the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
the success of peripheral intravenous catheter insertion | assessed up to 6 months
  Time until successful catheter placement

SECONDARY OUTCOMES:
patient satisfaction level scale | assessed up to 6 months
  Patient satisfaction levels with peripheral intravenous catheter placement procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No